CLINICAL TRIAL: NCT00631709
Title: REmote MOnitoring Transmission Evaluation of IPGs
Acronym: REMOTE-IPG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REMOTE-IPG 2008
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Pacemaker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Pacemaker Patients
  Interventions: Other: CareLink Remote Monitoring

INTERVENTIONS:
Other: CareLink Remote Monitoring — Substitution of CareLink Remote Monitoring of Pacemakers for in-clinic pacemaker follow-up visits

SUMMARY:
The purpose of this study is to evaluate the potential clinical and economic benefits of using CareLink remote management for pacemaker follow-up.

Study Objectives include:

1. To determine clinician perceived quality of care for CareLink remote follow-up.
2. To determine patient satisfaction with CareLink follow-up.
3. To estimate the time required to perform patient follow-up via CareLink remote transmissions.
4. To determine the percentage of regular CareLink follow-ups that do not require further in-clinic review of the patient.
5. To estimate potential patient cost avoidance for one year of follow up incorporating CareLink.
6. To evaluate compliance to scheduled CareLink transmissions with the remote management system

This is a non-randomized, multi-center, prospective study in which 120 patients who have a pacemaker are enrolled into the study and receive a CareLink monitor. Patients will replace their regularly scheduled pacemaker clinic follow-up visits with a CareLink remote transmission for 12months.

Patients will require a test transmission within 1 month after they receive their CareLink monitor. Afterwards, patients are followed via CareLink transmissions as per their usual clinic schedule for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a market released Medtronic pacemaker with automatic threshold management features for all active leads.
* Patients who have been implanted with their current pacemaker for at least 3 months.
* Patients who are willing, or who have caregivers willing, to use the Medtronic CareLink Monitor.
* Patients who are willing and able to sign an IRB/MEC approved patient informed consent.

Exclusion Criteria:

* Patients participating in another study that would affect the objectives of this study
* Patients who have already previously used a Medtronic CareLink Monitor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Southlake Regional Hospital, Newmarket, Ontario
  - CHUQ, L'Hotel Dieu de Quebec, Québec, Quebec